CLINICAL TRIAL: NCT00573664
Title: The Effectiveness and Safety of Gabapentin for Post-operative Pain After Cesarean Section: A Randomized Placebo-controlled Trial
Brief Title: The Effectiveness and Safety of Gabapentin for Post-operative Pain After Cesarean Section
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed a significant reduction in the pain scores
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose C.A. Carvalho, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-10; 07-0242-A
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Pain
Keywords: Cesarean section; Gabapentin
MeSH Terms: conditions — Pain | interventions — Gabapentin; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Gabapentin
  Interventions: Drug: Gabapentin
- 2 (Placebo Comparator): Placebo
  Interventions: Other: lactose

INTERVENTIONS:
Drug: Gabapentin — single oral dose of 600mg gabapentin
  Other Names: Neurontin
  Arms: 1
Other: lactose — Single dose
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether a single dose of gabapentin, given before cesarean section, will reduce pain in the initial 24 hours after surgery. Gabapentin has been very effective at treating pain after knee and hip operations, hysterectomies, and many other types of surgeries. We believe that it may be effective for treating pain after cesarean sections, but it has never been studied for this purpose.

DETAILED DESCRIPTION:
A cesarean section is a surgical procedure and, like all surgeries, there is pain after the operation. The purpose of this study is to find out if patients have less pain after a cesarean delivery when they receive a single dose of a gabapentin before the surgery. We are also interested in whether or not the dose of gabapentin reduces the need for other pain-killing medication during this time.

Patients will be randomly assigned to receive either gabapentin or a placebo. In addition, all patients will receive the usual standard of care and medication for pain (intrathecal morphine,oral paracetamol and diclofenac). At 4, 12, 24 and 48 hours after the operation, patients will be asked about their pain and satisfaction with pain management. The dose of gabapentin given is thought to be safe for the baby, and we plan to investigate whether the gabapentin has any effect on the baby's pain response when given his/her vitamin K injection. Gabapentin has also been shown to reduce long-term pain that can develop, and patients will be followed up at 6 weeks to be asked about their pain at that time.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective cesarean delivery

Exclusion Criteria:

* Patients unable to communicate in English
* Patients with an American Society of Anesthesiologists (ASA) classification of 3 or higher
* Patients with contraindications to any of the medications used in the study
* Patients with contraindications to spinal anesthesia
* Patients who have taken any pain medication in the past week
* Patients with fetuses having congenital abnormalities
* Patients with severe mental disorders
* Patients with HIV or hepatitis infections
* Intravenous drug users
* Patients with uncontrolled hypertension and diabetes
* Patients with central nervous system tumours

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Pain score by visual analogue scale (VAS) on movement at 24 hours postoperatively. | 24 hours

SECONDARY OUTCOMES:
Pain at rest and on movement by VAS at 4, 12, 24 & 48 hours postoperatively. | 48
Opioid consumption at 4, 12, 24 & 48 hours postoperatively. | 48
Assessment of sedation, pruritis, nausea, vomiting and dizziness on a 4-point scale (absent, mild, moderate, severe) and document treatment if required. | 48 hours
Time to first maternal request for supplemental analgesia. | 48 hours
Presence of pain 3 months postoperatively. | 3 months
Neonatal information: Apgar scores, arterial cord blood gases, arterial and venous cord blood gabapentin concentration, need for NICU admission | 48 hours
Neonatal pain response at vitamin K injection (0-100%) | 1 hour
Maternal gabapentin levels (25 patients) | 6 months (samples will be stored and sent together)

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada